CLINICAL TRIAL: NCT00902525
Title: Two Repeated Doses of Yttrium-90 Ibritumomab Tiuxetan (Zevalin®) as Salvage Treatment for Patients With Relapsed or Refractory Aggressive B-cell Lymphoma: a Phase II Study.
Brief Title: Zevalin Twice in Aggressive Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After enrolling 25 patients an interim analysis was done.The study was discontinued in the absence of the minimum number of 6 patients free of events
Sponsor: Gruppo Italiano Multiregionale per lo studio dei Linfomi e delle Leucemie (Other)
Collaborators: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZETAL07
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: two sequential doses of 90Y-Ibritumomab Tiuxetan
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 90Y-Ibritumomab Tiuxetan double dose (Experimental): 90Y-Ibritumomab Tiuxetan administered at 0.4 mCi/kg at phase 2 and then at 0.2 mCi/kg at phase 3
  Interventions: Drug: 90Y-Ibritumomab Tiuxetan

INTERVENTIONS:
Drug: 90Y-Ibritumomab Tiuxetan — All patients receive 2 courses of age-adjusted R-miniDHAP followed by two doses of 90Y-Ibritumomab Tiuxetan

SUMMARY:
Despite of the availability of treatment for this disease, this study is justified because no known therapies are really curative and it is necessary to look for new treatment options to improve the clinical outcome and prognosis of relapsed aggressive lymphoma. This study is designed for patients not eligible for high-dose chemotherapy and autologous stem cells transplantation.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the efficacy and safety of two sequential doses of 90Y-Ibritumomab Tiuxetan administered after salvage chemotherapy in patients with relapsed/refractory aggressive lymphoma non-eligible for HDC and ASCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75
2. Diagnosis of CD20+ B-diffuse large cell de novo or transformed or follicular lymphoma grade IIIb
3. Stage II, III, IV according to Ann Arbor criteria
4. Chemoresistant disease after first line treatment (CHOP-like + Rituximab) or relapsed patients after one or two lines of chemotherapy not-eligible for high dose chemotherapy and autologous stem cell transplantation
5. Performance status 0-2 according to WHO criteria
6. HIV negativity
7. Normal liver, lung and kidney function: conjugated bilirubin up to 2 x ULN, alkaline phosphatase and transaminases up to 2 x ULN, creatinine clearances ≥45 ml/min
8. Neutrophils count ³ 1.5 x 109/l, Haemoglobin ³ 9 g/dl, Platelets ³ 150 x 109/l and bone marrow involvement < 25% before first Zevalin infusion.
9. Neutrophils count ³ 1.5 x 109/l, Haemoglobin ³ 9 g/dl, Platelets ³ 100 x 109/l before second Zevalin infusion
10. Use of effective contraception for the entire treatment period in patients sexually active
11. Negative pregnancy test in child bearing potential women
12. Life expectancy > 6 months
13. Written informed consent

Exclusion Criteria:

1. More than two lines of prior chemotherapy before study entry
2. Prior high dose chemotherapy and autologous stem cell transplantation
3. HIV positivity
4. HBV positivity with the exception of patients with HBVcAb +, HbsAg -, HBs Ab+/- with HBV-DNA negative
5. HCV positivity with the exception of patients with no signs of active chronic hepatitis histologically confirmed
6. History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances
7. Uncontrolled diabetes (if receiving antidiabetic agents, subjects must be on a stable dose for at least 3 months before first dose of study drug
8. Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure (Attachment 5, NYHA Classification of Cardiac Disease), uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis
9. Pregnant or breastfeeding
10. CNS lymphoma involvement.
11. History of malignant carcinoma within the last 3 years other than squamous cell and basal cell carcinoma.
12. Cardiac failure with VEF < 40%
13. Clinical evidence of not controlled infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
An interim analysis on all the available data after the enrolment of the 15th patient (completion of the 1st stage) will be conducted, both for safety and efficacy. | after the enrolment of the 15th patient

SECONDARY OUTCOMES:
after the interim analysis, the writing committee of the study will evaluate to increase the second dose of Zevalin to 0.3 mCi/Kg. The same procedure will be applied to decide if the trial must be stopped after the enrolment of the 23rd patient. | after the enrolment of the 23rd patient

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Botto, MD, Study Director — SCDO Ematologia AOU San Giovanni Battista Torino; Umberto Vitolo, MD, Principal Investigator — SCDO Ematologia 2 AOU San Giovanni Battista Torino
Locations (12):
- Italy (12):
  - Divisione di Ematologia Ospedale SS Antonio e Biagio, Alessandria, AL
  - Istituto di Ematologia e Oncologia Medica L. Seragnoli Policlinco S. Orsola, Bologna, BO
  - Divisione di Ematologia, Spedali Civili, Brescia, BS
  - Divisione di Ematologia Ospedale Centrale di Bolzano, Bolzano, BZ
  - Divisione di Ematologia Ospedale Businco, Cagliari, CA
  - Divisione di Ematologia Ospedale Cardinale Panico, Tricase, LE
  - Divisione di Ematologia Ospedale Niguarda Cà Granda, Milan, MI
  - Divisione di Oncoematologia IRCC, Candiolo, TO
  - Divisione di Ematologia Istituto Nazionale Fondazione Pascale, Napoli
  - SC Ematologia Ospedale Maggiore Università Avogadro, Novara
  - Divisione di Oncoematologia Azienda Ospedalier S. Maria, Terni
  - SCDO Ematologia 2 AOU San Giovanni Battista, Turin